CLINICAL TRIAL: NCT03250533
Title: Analysis of the Effects of Phototherapy With Light-emitting Diodes (LED) and Electrical Stimulation in the Healing of Ulcers of Lower Diabetic Limbs: a Blind Controlled Randomized Clinical Test
Brief Title: Analysis of the Effects of LED Phototherapy and Electrical Stimulation in the Healing of Diabetic Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor, PT, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1143-0079
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Ulcer; Diabetes Mellitus
Keywords: Wound healing; Phototherapy; Electrotherapy
MeSH Terms: conditions — Ulcer; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Volunteers will also be randomized between groups:
  * LED treatment group 620 nm (G-LED 620; n = 13)
  * Treatment group with LED 940 nm (G-LED 940; n = 13)
  * Treatment group with fixed diphasic current (G-DF; n = 13)
  * Control group (G-C; n = 13)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LED 620 nm group (G-LED 620) (Experimental): The LED device in the red light spectrum, with a wavelength of 620 nm, will be applied over the full extent of the wound.
  Interventions: Device: Light emitting diodes (LED)
- LED 940 nm group (G-LED 940) (Experimental): The LED device in the infrared light spectrum, with a wavelength of 940 nm, will be applied over the full extent of the wound.
  Interventions: Device: Light emitting diodes (LED)
- Fixed diphasic current group (G-DF) (Experimental): The electrical stimulation will be carried out with the fixed diphasic current of the Dualpex 071 equipment, being applied throughout the extension of the wound.
  Interventions: Device: Fixed diphasic current
- Control group (G-C) (No Intervention): Volunteers from this group will not be submitted to treatment and will only be evaluated before, every 30 days, after the 12 week period and 30 days after the last evaluation. It is worth mentioning that, after the end of its participation, if the wound is not fully healed, the treatment will be offered with LED or diphasic current.

INTERVENTIONS:
Device: Light emitting diodes (LED) — The light-emitting diode (LED) device consists of a soft 15 x 15 cm blanket, which allows the body segment curvature of the cutaneous lesion to be monitored. The LEDs are fixed equidistant to obtain uniform irradiation over the entire ulcer. The wound site will be surrounded by a PVC film (polyvinyl chloride), to avoid contamination, for posterior positioning of the LED device, applying light directly and perpendicularly, with energy density of 6 J / cm². All LEDs will be calibrated prior to the start of applications in the Laboratory of Photobiophysics of the Faculty of Sciences and Letters of Ribeirão Preto, University of São Paulo, in which the wavelengths will be checked, the angle of radiation, power and power density.
  Arms: LED 620 nm group (G-LED 620); LED 940 nm group (G-LED 940)
Device: Fixed diphasic current — The electrical stimulation treatment will be performed with the fixed diphasic current of the Dualpex 071 equipment (Quark®, Piracicaba, SP, Brazil), with the monopolar technique, 100 Hz, maximum intensity of 1 mA / cm² of lesion for 10 minutes. Autoclave sterilized aluminum electrodes will be used, one on the lesion (negative pole) and the other transversal to the segment (positive pole). The size of the electrode will be proportional to the extension of the lesion, having as a means of contact between the electrode and the ulcer, sterile gauze moistened with 0.9% saline solution.
  Arms: Fixed diphasic current group (G-DF)

SUMMARY:
One of the important complications of DM is the diabetic foot that may present ulcers, which result from multiple risk factors, being diabetic peripheral neuropathy and ischemia due to peripheral vascular disease considered the main causes. In this way, the ulcers of the lower extremities of diabetics, have a complex and long cicatrization process. Faced with this, the treatment of chronic wounds is challenging, the diversity of treatments is great, however the search for new modalities of effective therapeutic resources, scientifically proven and financially feasible, that are available and easily accessible for clinical practice is still desirable . The aim of this study was to evaluate the responses of phototherapy with light emitting diodes (LED) and electrical stimulation with the fixed diphasic current (DF) in ulcers of diabetic patients. Diabetic volunteers who present with chronic skin ulcers will also be randomized (n = 13) to: Treatment group with LED 620 nm, Treatment group with LED 940 nm, Treatment group with fixed diphasic current and Control group. Interventions will occur three times a week for 12 weeks and evaluations will occur on the 1st, 30th, 60th, and 90th day of the intervention, followed by follow-up after 30 days of treatment completion.

DETAILED DESCRIPTION:
Background: Diabetes mellitus (DM) is a chronic disease currently considered a worldwide epidemic and has become a major public health problem. One of the important complications of DM is the diabetic foot that may present ulcers, which result from multiple risk factors, being diabetic peripheral neuropathy and ischemia due to peripheral vascular disease considered the main causes. In this way, the ulcers of the lower extremities of diabetics, have a complex and long healing process, as they present a reduction in the angiogenic response and deficiency of growth factors, making difficult the action of conventional treatments. The treatment of chronic wounds is challenging, the diversity of treatments is great, however the search for new modalities of effective, scientifically proven and financially viable therapeutic resources that are available and readily accessible to clinical practice is still desirable. Objective: To evaluate the responses of phototherapy with light emitting diodes (LED) and electrical stimulation with the fixed diphasic current (DF) in diabetic patient ulcers. METHODS: Diabetic volunteers of both genders, aged 30 to 65 years, who present chronic skin ulcers grade I or II will also be randomized (n = 13) in: Treatment group with LED 620 nm (G-LED 620) , Treatment group with LED 940 nm (G-LED 940), Treatment group with fixed diphasic current (G-DF) and Control group (GC). Interventions will occur three times a week for 12 weeks. The evaluations will take place on the pre-intervention day 1, 30, 60 and 90 days, followed by follow-up after 30 days of the end of the treatment, through the following instruments: numerical scale of pain, digital photography, infrared thermography, digital analgesimeter, Digital durometer, infrared plethysmography and bioimpedance. Statistical analysis: To analyze the data, normality test will be used to verify the distribution of the data and adequate statistical test for the appropriate inter- and intragroup comparisons, being thus considered two factors in the comparisons, time and group. A significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 30 to 65 years;
* Diabetic patients with neuropathic, ischemic or neuroischemic ulcers in the legs and / or feet;
* With a duration of 4 weeks or more;
* Being grade I and / or II lesions by the Meggitt-Wagner classification;
* Have a good degree of cognition evaluated by the Mini-Mental State Examination - MEEM (Brucki et al., 2003);
* Be under medical supervision and perform regular dressings and debridements of the wound.

Exclusion Criteria:

* Those presenting with an associated disease, such as renal, neurological, immunological, hematological or hepatic disease, which may interfere with evaluation and / or therapeutic procedures, and which are not related to diabetes;
* Malignancies (carcinomas);
* Use of medications that alter the healing process (corticosteroids, immunosuppressants, among others);
* Clinical signs of infection (sepsis), acute cellulitis, osteomyelitis or gangrene;
* Those who do not agree to sign the Free and Informed Consent Form;
* And who do not meet the inclusion criteria described.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of ulcer healing - Digital photography | Twelve weeks
  Percentage (%)

SECONDARY OUTCOMES:
Infrared thermography | Twelve weeks
  Skin temperature (Celsius Degree)
Numerical pain scale | Twelve weeks
  Intensity of pain (numerical scale)
Von frey digital analgesiometer | Twelve weeks
  Quantify the sensitivity
Digital Durometer | Twelve weeks
  Analyze the tissue firmness (Shore)
Infrared Plethysmography | Twelve weeks
  Changes in microvascular blood volume (mL/s)
Bioimpedance | Twelve weeks
  Phase angle (KHz)

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Guirro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Borges NCS, Soares LR, Perissini MM, Carvalho MS, Guirro ECO, Freitas MCF, Guirro RRJ. Photobiomodulation using red and infrared spectrum light emitting-diode (LED) for the healing of diabetic foot ulcers: a controlled randomized clinical trial. Lasers Med Sci. 2024 Oct 9;39(1):253. doi: 10.1007/s10103-024-04199-5. PMID 39382587